CLINICAL TRIAL: NCT02585908
Title: γδ T Cell Immunotherapy for Treatment of Gastric Cancer
Brief Title: Safety and Efficacy of γδ T Cell Against Gastric Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Doing Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Doing-001
Record Dates: First submitted 2015-10-22; First posted 2015-10-26 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-09

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental Group A(control group) (No Intervention): regular treatment and follow up
- Experimental Group B (Experimental): CIK will be used against tumor cells.
  Interventions: Biological: CIK
- Experimental Group C (Experimental): γδ T will be used against tumor cells.
  Interventions: Biological: γδ T
- Experimental Group D (Experimental): CIK and γδ T will be used against tumor cells.
  Interventions: Biological: CIK and γδ T

INTERVENTIONS:
Biological: CIK — CIK cells will be used against tumor cells.
  Arms: Experimental Group B
Biological: γδ T — γδ T cells will be used against tumor cells.
  Arms: Experimental Group C
Biological: CIK and γδ T — CIK and γδ T cells will be used against tumor cells.
  Arms: Experimental Group D

SUMMARY:
In this study, safety and effects of γδT cells on human gastric cancer are going to be investigated.

DETAILED DESCRIPTION:
PBMC of the patient will be separated from peripheral blood. After making them potential cancer killer γδ T Cell and CIK, they will be infused to the patients as immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age:30-75
2. Karnofsky performance status >50
3. Diagnosis with gastric cancer based on histology or the current accepted radiological measures.
4. Classification tumor,nodes,metastasis-classification(TNM) stage: Ⅱ,Ⅲ,Ⅳ
5. Patients who have a life expectancy of at least 12 weeks
6. Ability to understand the study protocol and a willingness to sign a written informed consent document

Exclusion Criteria:

1. Any significant medical or psychiatric illness that would prevent the patient from giving informed consent or from following the study procedures.
2. Known human immunodeficiency virus (HIV) infection.
3. Active and/or severe infection (e.g. tuberculosis, sepsis and opportunistic infections, active hepatitis B virus (HBV) or active hepatitis C virus (HCV) infection).
4. Other serious underlying medical conditions, which, in the Investigator's judgment, could impair the ability of the patient.
5. Pregnancy

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Reduced size of the tumor. | up to one year
  Tumor load will be evaluated by RECIST criteria.

SECONDARY OUTCOMES:
Safety, as measured by the rate of adverse events and serious adverse events | up to two years
  Safety, as measured by the rate of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: li gangyi, master, Study Chair — Beijing Doing Biomedical Co., Ltd.
Locations (4):
- China (4):
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Huai'An First People'S Hospital, Huaian, Jiangsu
  - Hangzhou Cancer Hospital, Hangzhou, Zhejiang